CLINICAL TRIAL: NCT03847662
Title: Scaling up Small-Scale Food Processing: A Strategy to Promote Food Security Among Women Subsistence Farmers in Rural Vietnam
Brief Title: Scaling up Small-Scale Food Processing to Promote Food Security Among Women Farmers in Rural Vietnam
Status: Completed | Type: Observational
Sponsor: National Institute of Nutrition, Vietnam (Other Government)
Collaborators: Toronto Metropolitan University (Other); Global Affairs Canada (Other); International Development Research Centre, Canada (Other Government)
Responsible Party: Principal Investigator, Nguyen Do Huy, Principle Investigator, National Institute of Nutrition, Vietnam
Other Study IDs: CIFSRF 108124
Record Dates: First submitted 2018-11-07; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Food Insecurity; Stunting; Wasting; Underweight; Anemia
Keywords: Food Insecurity; Stunting; Wasting; Underweight; Anemia; Complimentary Foods; Food Fortification; Complimentary Feeding
MeSH Terms: conditions — Growth Disorders; Cachexia; Thinness; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community Based Production and Access of Complimentary Foods: Nine communes were randomly selected with the cluster inclusion criteria as having high levels of; agricultural production, childhood under-nutrition and food security. This was carried out in the three rural mountainous provinces of Lao Cai, Lai Chau, and Ha Giang. In each of these provinces, one district and three subsequent communes were selected, for a total of 9 communes. The districts of Bat Xat, Tam Duong, and Vi Xuyen were selected in Lao Cai, Lai Chau and Ha Giang province respectively. This second stage district sampling selected sites with similar characteristic of population density, area, number of women of reproductive age(15-35y), percentage of children(<2y), income primarily from agricultural production, poverty and climate data.
  Changes were observed on food security and nutritional status with exposure to community based self reported purchasing local agricultural products and access to locally produced fortified complimentary foods.

SUMMARY:
This repeated measures, cluster randomized, cohort trial design was carried out in three provinces in the northern mountainous area of Vietnam. Communes here were randomly selected for community based interventions with local production complimentary foods and marketing and distribution of fortified complimentary foods.

DETAILED DESCRIPTION:
In rural northern Vietnam, childhood stunting rates are high. In Lào Cai province, female subsistence farmers grow crops, but face barriers sending produce to markets. The present intervention purchases local crops from local women subsistence farmers which are processed in local small-scale food processing facilities to produce instant fortified complementary foods for weaning.

Methods: A repeated measures survey was conducted from October to November 2016, with Caregiver-Child(<2y) pairs (n=800) in the provinces of Lai Chau, Lao Cai and Ha Giang. Anthropometric data of mother/child dyads was assessed and logistic regression analysis of stunted and underweight children explored associated factors. These included: core infant and young child feeding practices indicators, food insecurity, antenatal care check-ups, core water/sanitation, anemia and hygiene indicators.

This project leveraged the experience of the National Institute of Nutrition of Vietnam to ensure HACCP standards during manufacture. Locally grown rice was combined with a Zn/Fe premix before extrusion and hammer-milling. Local vegetables such as: "Sweet leaf" (Sauropus androgynous), pumpkin, Shiitake mushrooms (Lentinula edodes) and carrots were made into complimentary foods and sold locally.

ELIGIBILITY:
Inclusion Criteria:

* Child participants must be younger than 2y at baseline.
* Caregivers must volunteer and were required to give informed written consent

Exclusion Criteria:

* Free from oedema
* Free from physical and mental disabilities
* Free from memory disorders and/or mental illness

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Perspective participants from these 9 communes, were invited to participate based on the inclusion criteria of the project and randomization lists will be made from the lists of children (< 2y) from the commune health centers. From these lists, 800 children will be randomly selected and categorized by age into different groups: 100 infants of 0-5 months, 400 infants of 6-12 months, and 200 children of 12-23 months will be selected.
  A initial cross-sectional Baseline survey with a was conducted from October to November 2016, with Caregiver-Child(<2y) pairs (n=799) in the provinces of Lai Chau, Lao Cai and Ha Giang.
Sampling Method: Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Household Food Insecurity Access Scale | Nov 2016-June 2018
  Score from 1-27 indicating household food Insecurity. Where higher scores indicate greater food insecurity. This was taken at the beginning of intervention in Nov 2016 till completion in June 2018.

SECONDARY OUTCOMES:
Weight in kilograms | Nov 2016-June 2018
  Stunting (Height-for-age Z score <-2SD), Underweight (Weight-for-age Z score<-2SD), Wasting (Weight-for-height Z score<-2SD) compared with World Health Organization's growth charts.
Height in Meters | Nov 2016-June 2018
  Stunting (Height-for-age Z score <-2SD), Underweight (Weight-for-age Z score<-2SD), Wasting (Weight-for-height Z score<-2SD) compared with World Health Organization's growth charts.
Age in Months | Nov 2016-June 2018
  Stunting (Height-for-age Z score <-2SD), Underweight (Weight-for-age Z score<-2SD), Wasting (Weight-for-height Z score<-2SD) compared with World Health Organization's growth charts.
Hemoglobin Levels of Children (<2y) | Nov 2016-June 2018
  Hemoglobin levels among Children participants assessed by finger prick blood sampling.

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data available.

REFERENCES:
- See also: Video Overview of the Project (CIFSRF 108124) — https://www.youtube.com/watch?v=NrRq9SRB9dk
- See also: CIFSRF report — https://www.idrc.ca/en/project/scaling-small-scale-food-processing-therapeutic-and-complementary-foods-children-vietnam